CLINICAL TRIAL: NCT06590155
Title: Role of Erythropoietin in Neonates With Hypoxic Ischemic Encephalopathy
Brief Title: Erythropoietin in HIE Neonate
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Saber Fahmy, resident doctor at internal medicine department, Assiut University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Erythropoietin in HIE neonate
Record Dates: First submitted 2024-02-24; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neonatal Hypoxic Ischemic Encephalopathy
MeSH Terms: interventions — Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- to delineate the role of erythropoietin in improving neonatal hypoxic ischemic encephalopathy (Experimental): Erythropoietin was administered in the first weeks of life at different multiple doses between 259-1000 UI/KG/D for 3 days
  Interventions: Drug: Erythropoietin
- Role of Erythropoietin in neonate hypoxic ishemic encephalopathy (Other): EPO reduces the need for blood transfusions in premature infants. To cross the blood-brain barrier
  Interventions: Drug: Erythropoietin
- Role of Erythropoietin in neonatal hypoxic ischemic encephalopathy (No Intervention): prevent apoptosis of erythroid progenitor cells and to enhance their maturation and proliferation

INTERVENTIONS:
Drug: Erythropoietin — the role of erythropoietin in improving neonatal hypoxic ischemic encephalopathy
  Arms: Role of Erythropoietin in neonate hypoxic ishemic encephalopathy; to delineate the role of erythropoietin in improving neonatal hypoxic ischemic encephalopathy

SUMMARY:
this study is aim to delineate the role of erythropoietin in improving neonatal hypoxic ischemic encephalopathy the study is conducted to answer the question : is erythropoietin will improve neonatal hypoxic ischemic encephalopathy?

DETAILED DESCRIPTION:
Hypoxic-ischemic encephalopathy (HIE) remains a major cause of morbidity and mortality. HIE causes 23% of neonatal deaths . Erythropoietin is a 34kDa glycoprotein that was originally identified because of its role in erythropoiesis. In the fetus, EPO is produced in the liver, and, following the neonatal period, EPO is produced in the kidney and the liver. EPO is a cytokine with pleiotropic functions including erythropoiesis, modulation of inflammatory and immune responses. EPO and the EPO receptor (EPO-R) are expressed by a variety of cell types in the brain including neuronal progenitor cells. EPO transport across the blood-brain barrier is limited by its large size. Only 1% to 2% of circulating EPO crosses the blood-brain barrier under normal circumstances, most likely via passive diffusion . EPO provides a mechanism to maintain or re-establish the function of all other cells in challenging physiological conditions (e.g., hypoxia) . EPO's main role is to prevent apoptosis of erythroid progenitor cells and to enhance their maturation and proliferation . The use of EPO reduces the need for blood transfusions in premature infants. To cross the blood-brain barrier, high doses at 2000 to 5000 IU/kg body weight are administered either early or late for prolonged periods of time. These high doses are well tolerated in preterm infants (i.e., EPO is safe and devoid of untoward complications in this context . In previos studies , The first dose of r-Hu-EPO was administered at 1 to 48 h after birth, followed by doses every other day for 2 weeks. At 18 months-of-age neurodevelopmental outcomes were assessed. Improved long-term outcomes in the r-Hu-EPO-treated infants were evident after moderate HIE, but not in those with severe HIE. There were no side-effects from r-HuEPO treatment .

ELIGIBILITY:
Inclusion Criteria:

- neonates who less than 1 month suffer from hypoxic ischemic encephalopathy

Exclusion Criteria:

* neonates who more than 1 month
* neonates who suffer from brain insults other than HIE

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Estimated)
Dates: Start 2024-11-24 (Estimated); Primary Completion 2029-02-24 (Estimated); Study Completion 2029-02-24 (Estimated)

PRIMARY OUTCOMES:
oxygen saturation in neonates hypoxic ischemic encephalopathy after treatment byerythropoietin | Baseline
  EPO provides a mechanism to maintain or re-establish the function of all other cells in challenging physiological conditions e.g., hypoxia

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university children hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Erythropoietin: a novel therapy for hypoxic-ischaemic encephalopathy — https://www.frontiersin.org/articles/10.3389/fped.2022.1074287/full
- See also: Erythropoietin in perinatal hypoxic-ischemic — https://www.degruyter.com/document/doi/10.1515/jpm-2018-0360/html